CLINICAL TRIAL: NCT01001728
Title: A Randomised Trial Investigating the Prone Treatment Position as a Method of Sparing Healthy Tissues in Women Prescribed Breast Radiotherapy (SuPr Study)
Brief Title: SuPr Study (Supine Versus Prone Treatment Position in Breast Radiotherapy)
Acronym: SuPr
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCR3131
Record Dates: First submitted 2009-10-26; First posted 2009-10-27 (Estimated); Last update posted 2016-05-23 (Estimated); Status verified 2016-05

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Radiotherapy; Prone position
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prone Position (Active Comparator): Patients will lie on their fronts on an in-house designed board comprising an arm positioning device registerable to the couch-top, together with a styrofoam/ memory foam mattress. The ipsilateral breast will drop through an aperture in the mattress. The distance from the nipple to the superior, inferior and lateral aspects of the aperture will be recorded along with the distance of the nipple from the couch-top. Arms will be extended as far as possible above the head and the position of the arm immobilisation handles recorded. The head will be turned to the contralateral side. The contralateral breast will be pulled laterally such that it is as flat as possible beneath the patient. Measurements will be taken in order to relate the position of the bi-lateral tattoos to the orthogonal lasers. A fourth tattoo will be marked on the patient's back in line with the A-P laser. The position will be reproduced at treatment using measurements from the tattoo to the laser.
  Interventions: Radiation: Imaging investigations (with radiation)
- Supine position (Active Comparator): For the supine position, patients will be positioned on a customized supine breast board co-registerable to the couch-top to CT and the treatment machines. Arms will be placed above the head in supports. Arm and head position will be recorded along with the angle of the board (which is adjusted such that the sternum is parallel to the couch-top). Tattoos will be marked bi-laterally and medially in a defined relationship to orthogonal lasers. The position will be reproduced at treatment using the above measurements, tattoos and lasers.
  Interventions: Radiation: Imaging investigations (with radiation)

INTERVENTIONS:
Radiation: Imaging investigations (with radiation)

SUMMARY:
A randomised, two-arm, non-blinded crossover study investigating the impact of treatment position (prone versus supine) upon reproducibility of tumour bed position in patients undergoing breast radiotherapy following excision of early breast cancer.

DETAILED DESCRIPTION:
To establish whether or not the prone (face down) position reduces exposure of healthy tissue to radiation when compared to the supine position. To compare patient comfort and acceptability in each of the prone and supine positions. To perform a time and motion study for radiotherapy planned and delivered in each of the prone and supine positions.

ELIGIBILITY:
Inclusion Criteria:

* Complete microscopic excision of early stage invasive ductal or lobular carcinoma (pT1-3b N0-1 M0) with breast preservation.
* Paired titanium clips marking anterior, posterior, and radial walls of excision cavity
* Breast cup size C or above
* Recommendation for whole breast radiotherapy
* No requirement for nodal irradiation
* Ability to lie prone on breast board
* For left-sided breast cancer patients, cardiac and LAD doses must be ≤10% greater than those predicted for the supine position.
* For all patients, the following absolute dose constraints should be met: ≤5% of heart volume to receive 18Gy and ≤10% of ipsilateral lung volume to receive ≥20Gy
* Age ≥18
* PS ≤1
* No previous radiotherapy to the affected breast
* No concomitant herceptin
* Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule.
* Written informed consent given according to ICH/GCP before registration/ randomisation.
* Patients can only be randomised into this trial once.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2008-11; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Interfraction reproducibility of tumour bed position (Reproducibility of tumour bed position in supine versus prone positions compared using the difference in mean daily displacement in tumour bed centre of gravity over a course of radiotherapy in 3D). | End of radiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Professor John Yarnold, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- Royal Marsden NHS Foundation Trust, Sutton, Surrey, United Kingdom